CLINICAL TRIAL: NCT03524729
Title: Do Rocker Bottom Shoes and Ankle-Foot Orthoses Reduce Pain and Improve Mobility for Ankle Osteoarthritis Patients?
Brief Title: Do Rocker Bottom Shoes and Ankle-Foot Orthoses Reduce Pain and Improve Mobility for Ankle Osteoarthritis Patients
Acronym: RB/AFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F2278-R; RX002278 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2018-03-29; First posted 2018-05-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Ankle Osteoarthritis; Healthy Ankles
Keywords: Rocker bottom shoe; Ankle-foot orthosis; Ankle osteoarthritis

STUDY DESIGN:
Intervention Model Description: The osteoarthritis participants will wear the control shoe, rocker bottom shoe, and AFO for multiple weeks each. The order of the treatments (control shoe, rocker bottom shoe, and AFO) will be randomize.
  The control group will only wear the control shoe.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ankle osteoarthritis patients (Active Comparator): Ambulatory adult patients (18+) with ankle osteoarthritis.
  Interventions: Device: Rocker bottom shoe; Device: Ankle foot orthosis; Device: Standard walking shoe
- Healthy control subjects (Other): Ambulatory adults (18+) with no known ankle osteoarthritis.
  Interventions: Device: Standard walking shoe

INTERVENTIONS:
Device: Rocker bottom shoe — Walking shoe with a anterior posterior rocker sole.
  Arms: Ankle osteoarthritis patients
Device: Ankle foot orthosis — Dynamic carbon fiber ankle brace.
  Arms: Ankle osteoarthritis patients
Device: Standard walking shoe — Standard walking shoe (control shoe) with no rocker sole.

SUMMARY:
Ankle osteoarthritis (OA) is a painful, progressive condition that can severely limit physical activity and reduce quality of life. Rocker bottom (RB) shoes and ankle-foot orthoses (AFOs) are commonly used as non-surgical treatments for ankle OA. RB shoes have a curved sole in the toe to heel direction that may alleviate joint pain by reducing ankle range of motion (ROM). Similarly, AFOs may reduce joint motion by securing the foot and ankle within the ankle-foot orthosis (AFO) frame. This study aims to determine the ability of RB shoes and AFOs to improve mobility, by relieving pain and reducing joint ROM.

DETAILED DESCRIPTION:
The investigators' objective is to compare two non-surgical treatments (RB shoes and Toeoff brand AFOs) in OA subjects by measuring their mobility and pain during and after a multi-week trial period. The investigators will use a biplane fluoroscopy system to measure foot joint motion for each condition (RB shoe, AFO, control shoe). This will yield clinical and biomechanical measures of the effect of each orthotic on mobility, pain, and joint ROM in an ankle OA population. The investigators will also compare the clinical and biomechanics outcomes of OA subjects to those of control subjects. This information will provide evidence to support clinical decision making.

Aim 1: Compare the daily sep count, self-selected walking speed, clinical outcome measures (PROMIS surveys) of a control shoe, RB shoe, and AFO worn over a multi-week trial period.

Aim 2: Evaluate the effect of a control shoe, RB shoe, and AFO on the foot and ankle joints range of motion.

Aim 3: Compare the ankle OA clinical and biomechanical outcome measures for the control shoe, RB shoe, and AFO to a healthy control group wearing control shoes.

The efficacy of conservative treatments such as RB shoes and AFOs for managing OA pain and discomfort is not well supported by clinical evidence. By using biplane fluoroscopy along with validated clinical measures of pain and mobility, this study will elucidate the mechanism by which RB shoes and AFOs biomechanically alter foot and ankle function. Identifying beneficial treatment strategies for people with ankle OA will help them regain their mobility and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

For osteoarthritis patients:

* radiographic evidence of tibiotalar osteoarthritis
* ambulatory

For healthy controls:

* ambulatory
* aged 18 or older

Exclusion Criteria:

For osteoarthritis patients and healthy controls:

* subtalar joint arthritis
* plans for surgical treatment of ankle osteoarthritis within the next 4 months
* surgical, neurological, metabolic, or lower limb musculoskeletal problem that would impair study measures
* inability to walk unassisted during short, repeated walking trials
* rheumatoid arthritis
* inadequate cognitive or language function to consent or to participate
* no phone number or stable mailing address

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J. Sangeorzan, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected will be de-identified and placed in publically accessible online data repositories.
Time Frame: Data will be posted ad-hoc on an ongoing basis.
Access Criteria: Once posted, the data is available to the public.

RESULTS

PARTICIPANT FLOW:
Groups:
- Ankle Osteoarthritis Patients: AFO, Then RB, Then C; Ankle Osteoarthritis Patients: C, Then RB, Then AFO; Ankle Osteoarthritis Patients: C, Then AFO, Then RB; Ankle Osteoarthritis Patients: RB, Then C, the AFO; Ankle Osteoarthritis Patients: RB, the AFO, Then C: Ambulatory adult patients (18+) with ankle osteoarthritis. Rocker bottom shoe (RB): Walking shoe with a anterior posterior rocker sole. Ankle foot orthosis (AFO): Dynamic carbon fiber ankle brace. Control (C): Standard walking shoe (control shoe) with no rocker sole.
  First Intervention (3 weeks) Washout (1 week) Second Intervention (3 weeks) Washout (1 week) Third Intervention (3 weeks)
Period: Overall Study
Arm/Group | Ankle Osteoarthritis Patients: AFO, Then RB, Then C | Healthy Control Subjects | Ankle Osteoarthritis Patients: C, Then RB, Then AFO | Ankle Osteoarthritis Patients: C, Then AFO, Then RB | Ankle Osteoarthritis Patients: RB, Then C, the AFO | Ankle Osteoarthritis Patients: RB, the AFO, Then C
Started | 2 | 1 | 2 | 2 | 2 | 2
Completed | 2 | 1 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects | Total
Number analyzed (Participants) | 10 | 1 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 7 | 0 | 7
Age, Continuous [Mean (Full Range); unit: years] | 66 [56 to 75] | 62 [62 to 62] | 65 [56 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 1 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Daily Step Count (# Steps)
Description: The daily step count of a participant as measured by a body worn pedometer.
Time Frame: Three weeks
Population: numbers analyzed are different as there was issue with the data collection device and data were not recorded
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Ankle Osteoarthritis Patients: AFO, Then RB, Then C | Healthy Control Subjects | Ankle Osteoarthritis Patients: C, Then RB, Then AFO | Ankle Osteoarthritis Patients: C, Then AFO, Then RB | Ankle Osteoarthritis Patients: RB, Then C, the AFO | Ankle Osteoarthritis Patients: RB, the AFO, Then C
Number analyzed (Participants) | 2 | 0 | 2 | 1 | 2 | 1
steps
  with C: number analyzed (Participants) | 2 | 0 | 2 | 0 | 0 | 1
  with C | 3453 (244) |  | 2399 (268) |  |  | 3453 (NA) — no standard deviation for 1 participant
  With AFO: number analyzed (Participants) | 2 | 0 | 2 | 1 | 1 | 1
  With AFO | 2745 (1613) |  | 933 (671) | 2043 (NA) — no standard deviation for 1 participant | 503 (NA) — data were not recorded, issue with data collection device for 1 participant. therefore no SD | 2745 (NA) — no standard deviation for 1 participant
  With RB: number analyzed (Participants) | 2 | 0 | 2 | 0 | 0 | 1
  With RB | 2053 (776) |  | 2574 (82) |  |  | 2053 (NA) — no standard deviation for 1 participant

2. Secondary Outcome: Ankle Joint Range of Motion (Degrees)
Description: Range of motion of the ankle joint in degrees as measured by biplane fluoroscopy and/ or CT scan
Time Frame: Three weeks
Population: Due to COVID-19 delays and moving to a remote data collection, the investigators were unable to capture this outcome measure data
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Self-selected Walking Speed
Description: Self-selected walking speed as measured with a stop watch when walking a fixed distance.
Time Frame: Three weeks
Population: as for outcome 2
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Qualitative Assessment of Patient Device Wearing
Description: Would you continue to wear the device if you were not part of the study? Why/why not?
Time Frame: Three weeks
Population: as for outcome 2
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function
Description: Self reported capability of physical function Min: 0 Max: 100 A higher score indicates better physical function
Time Frame: three weeks
Population: numbers analyzed are different as there was issue with the data collection device and data were not recorded
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Osteoarthritis Patients: AFO, Then RB, Then C | Healthy Control Subjects | Ankle Osteoarthritis Patients: C, Then RB, Then AFO | Ankle Osteoarthritis Patients: C, Then AFO, Then RB | Ankle Osteoarthritis Patients: RB, Then C, the AFO | Ankle Osteoarthritis Patients: RB, the AFO, Then C
Number analyzed (Participants) | 2 | 0 | 2 | 1 | 1 | 1
score on a scale
  C | 50.9 (8.7) |  | 37.3 (7.7) | 37.9 (NA) — only one participant, therefor no SD | 43.5 (NA) — only one participant, therefor no SD | 50.9 (NA) — only one participant, therefor no SD
  AFO | 52 (5.1) |  | 22.5 (7.4) | 41 (NA) — only one participant, therefor no SD | 45.6 (NA) — only one participant, therefor no SD | 52 (NA) — only one participant, therefor no SD
  RB | 50.35 (2.2) |  | 41.4 (26.3) | 41.6 (NA) — only one participant, therefor no SD | 45.6 (NA) — only one participant, therefor no SD | 50 (NA) — only one participant, therefor no SD

6. Secondary Outcome: Fast Walking Speed
Description: Fast walking speed as measured with a stop watch when walking a fixed distance.
Time Frame: Three weeks
Population: as for outcome 2
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Timed-up-and-go
Description: Self-selected walking speed get out of a chair, walk to a line, turn around, walk back to the chair and sit down as measured with a stop watch.
Time Frame: Three weeks
Population: as for outcome 2
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Qualitative Assessment of Patient Satisfaction With the Device
Description: Do you like the device? Why/why not?
Time Frame: Three weeks
Population: as for outcome 2
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Qualitative Assessment of Device Preference
Description: Do you have a preference to one of the treatments? Which one? Why/why not?
Time Frame: Three Months
Population: as for outcome 2
Arm/Group | Ankle Osteoarthritis Patients | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference
Description: Self reported consequences of pain on relevant aspects of one's life.
  Min:0 Max: 100 A higher score indicates more pain interference
Time Frame: three weeks
Population: issue with data collection device, data were not collected for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Osteoarthritis Patients: AFO, Then RB, Then C | Healthy Control Subjects | Ankle Osteoarthritis Patients: C, Then RB, Then AFO | Ankle Osteoarthritis Patients: C, Then AFO, Then RB | Ankle Osteoarthritis Patients: RB, Then C, the AFO | Ankle Osteoarthritis Patients: RB, the AFO, Then C
Number analyzed (Participants) | 2 | 0 | 2 | 1 | 1 | 1
score on a scale
  C | 54 (2.8) |  | 56 (14.7) | 61 (NA) — only one participant, therefor no SD | 61 (NA) — only one participant, therefor no SD | 54 (NA) — only one participant, therefor no SD
  AFO | 52 (2.2) |  | 22 (4.3) | 41 (NA) — only one participant, therefor no SD | 45 (NA) — only one participant, therefor no SD | 52 (NA) — only one participant, therefor no SD
  RB | 50 (2.6) |  | 41 (1) | 42 (NA) — only one participant, therefor no SD | 46 (NA) — only one participant, therefor no SD | 50 (NA) — only one participant, therefor no SD

11. Secondary Outcome: Foot and Ankle Ability Measure (FAAM)
Description: American Academy of Orthopaedic Surgeons Foot and Ankle Module questionnaire designed to assess foot and ankle conditions.
  Min:0 Max: 100 Higher= better
Time Frame: three weeks
Population: issue with data collection device, data were not collected for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Osteoarthritis Patients: AFO, Then RB, Then C | Healthy Control Subjects | Ankle Osteoarthritis Patients: C, Then RB, Then AFO | Ankle Osteoarthritis Patients: C, Then AFO, Then RB | Ankle Osteoarthritis Patients: RB, Then C, the AFO | Ankle Osteoarthritis Patients: RB, the AFO, Then C
Number analyzed (Participants) | 2 | 0 | 2 | 1 | 1 | 1
score on a scale
  C | 71 (23) |  | 70 (35) | 45 (NA) — only 1 participant, no SD | 50 (NA) — only 1 participant, no SD | 72 (NA) — only 1 participant, no SD
  AFO | 92 (1) |  | 63 (26) | 57 (NA) — only 1 participant, no SD | 30 (NA) — only 1 participant, no SD | 92 (NA) — only 1 participant, no SD
  RB | 70 (42) |  | 60 (7) | 64 (NA) — only 1 participant, no SD | 51 (NA) — only 1 participant, no SD | 70 (NA) — only 1 participant, no SD

12. Secondary Outcome: Numeric Pain Rating Scale
Description: The Numeric Pain Rating Scale is a measure of pain intensity in adults in which the respondent selects a whole number (0-10) that best reflects the intensity of her / his pain. The scale will be administered verbally.
  scale of 1-10 higher= worse
Time Frame: three weeks
Population: issue with data collection device, data were not collected for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Osteoarthritis Patients: AFO, Then RB, Then C | Healthy Control Subjects | Ankle Osteoarthritis Patients: C, Then RB, Then AFO | Ankle Osteoarthritis Patients: C, Then AFO, Then RB | Ankle Osteoarthritis Patients: RB, Then C, the AFO | Ankle Osteoarthritis Patients: RB, the AFO, Then C
Number analyzed (Participants) | 2 | 0 | 2 | 1 | 1 | 1
score on a scale
  C | 3.5 (2.1) |  | 5 (2.8) | 5 (NA) — only 1 participant, no SD | 2 (NA) — only 1 participant, no SD | 3.5 (NA) — only 1 participant, no SD
  AFO | 3 (1.4) |  | 3.5 (4.9) | 5 (NA) — only 1 participant, no SD | 5 (NA) — only 1 participant, no SD | 3 (NA) — only 1 participant, no SD
  RB | 2.5 (0.7) |  | 3 (4.2) | 6 (NA) — only 1 participant, no SD | 7 (NA) — only 1 participant, no SD | 2.5 (NA) — only 1 participant, no SD

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: we did not expect mortality during this study
Groups:
- Ankle Foot Orthosis (AFO): Ankle foot orthosis (AFO): Dynamic carbon fiber ankle brace.
- Rocker Bottom Shoe (RB): Rocker bottom shoe (RB): Walking shoe with a anterior posterior rocker sole.
- Control (C): Control (C): Standard walking shoe (control shoe) with no rocker sole.
Arm/Group | Ankle Foot Orthosis (AFO) | Healthy Control Subjects | Rocker Bottom Shoe (RB) | Control (C)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/1 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/1 | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/1 | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ankle Foot Orthosis (AFO) (N=8) | Healthy Control Subjects (N=1) | Rocker Bottom Shoe (RB) (N=8) | Control (C) (N=8)
infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03524729/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT03524729/ICF_001.pdf